CLINICAL TRIAL: NCT01965262
Title: A Clinical Assessment of the Hemacopolymer Daily Disposable Limbal Ring Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CV13-545
Record Dates: First submitted 2013-10-11; First posted 2013-10-18 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hema-copolymer Lens (Active Comparator): Participants were randomized to wear the Hema-copolymer lens pair for one week during the cross over study.
  Interventions: Device: Hema-copolymer Lens; Device: etafilcon A Lens
- etafilcon A Lens (Active Comparator): Participants were randomized to wear the etafilcon A lens pair for one week during the cross over study.
  Interventions: Device: Hema-copolymer Lens; Device: etafilcon A Lens

INTERVENTIONS:
Device: Hema-copolymer Lens — contact lens
Device: etafilcon A Lens — contact lens

SUMMARY:
This purpose of this study is to compare the clinical performance and subjective acceptance of two different daily disposable limbal ring lenses.

DETAILED DESCRIPTION:
This is a subject-masked, dispensing study designed to evaluate the clinical performance and subjective acceptance when comparing two different daily disposable limbal ring lenses. Limbal ring lenses, which as well as correcting vision, have a colored ring which enhance the wearer's iris and are particularly popular in East Asian countries.

ELIGIBILITY:
Inclusion Criteria:

Subjects will only be eligible for the study if:

* They are 18 years of age and above.
* They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
* They are willing and able to follow the protocol.
* They agree not to participate in other clinical research for the duration of this study.
* They can attain at least 6/9 in each eye with the study lenses within the available power range.
* They can be fitted with study lenses within the available power range.
* The currently use soft contact lenses, or have done so within the last six months.

Exclusion Criteria:

Subjects will not be able to take part in the study if:

* They have an ocular disorder which would normally contraindicate contact lens wear.
* They have a systemic disorder which would normally contraindicate contact lens wear.
* They are using any topical medication such as eye drops or ointment.
* They have had cataract surgery.
* They have had corneal refractive surgery.
* They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
* They are pregnant or lactating.
* They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
* They have any infectious disease which would normally contraindicate contact lens wear, or may, in the opinion of the investigator, pose a risk to study personnel; or any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reactions.
* They have taken part in any other clinical trial or research, within two weeks prior to starting this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carole Maldonado-Codinal, PhD, Principal Investigator — Eurolens Research
Locations (1):
- Eurolens Research - The University of Manchester, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty subjects were dispensed lenses, and nineteen subjects successfully wore both study products.
Groups:
- Hema-copolymer Lens, Then Etafilcon A Lens: Participants were randomized to wear the Hema-copolymer lens pair for one week then cross over to the etafilcon A lens pair.
- Etafilcon A Lens, Then Hema-copoloymer Lens: Participants were randomized to wear the etafilcon A lens pair for one week then cross over to the Hema-copolymer lens lens pair.
Period: First Intervention (7 Days)
Arm/Group | Hema-copolymer Lens, Then Etafilcon A Lens | Etafilcon A Lens, Then Hema-copoloymer Lens
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention (7 Days)
Arm/Group | Hema-copolymer Lens, Then Etafilcon A Lens | Etafilcon A Lens, Then Hema-copoloymer Lens
Started | 15 | 15
Completed | 14 | 5
Not Completed | 1 | 10
Not completed — Discontinued | 0 | 1
Not completed — Poor lens fit | 0 | 9
Not completed — Poor visual acuity | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Baseline Characteristics: Randomized to wear the Hema-copolymer lens pair or the etafilcon A lens pair for one week then cross over to the alternate pair
  Hema-copolymer Lens: Hema-copolymer lens pair or the Etafilcon A lens pair
  etafilcon A Lens: Hema-copolymer lens pair or the Etafilcon A lens pair
Arm/Group | Overall Baseline Characteristics
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (11.2)
Age, Continuous [Mean (Full Range); unit: years] | 29.2 [18 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity - Hema-copolymer and Etafilcon A
Description: Visual acuity measured by logMAR of hema-copolymer and etafilcon A lenses assessed at baseline.
Time Frame: Baseline
Population: All 30 subjects were dispensed lenses, and visual acuity measurements were obtained at baseline.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Hema-copolymer Lens: Participants were randomized to wear the Hema-copolymer lens pair for one week during the cross over study.
  Hema-copolymer: contact lens
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 30 | 30
logMAR
  High Contrast | -0.08 (0.09) | -0.04 (0.09)
  Low Contrast | 0.17 (0.10) | 0.20 (0.14)

2. Primary Outcome: Visual Acuity - Hema-copolymer and Etafilcon A
Description: Visual acuity measured by logMAR for hema-copolymer and etafilcon A lenses assessed at 1 week.
Time Frame: 1 week
Population: 11 subjects discontinued the study. Missing data of 1 subject for hema-copolymer group.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 28 | 20
logMAR
  High Contrast | -0.08 (0.10) | -0.04 (0.10)
  Low Contrast | 0.18 (0.09) | 0.23 (0.10)

3. Primary Outcome: Biomicroscopy - Hema-copolymer and Etafilcon A
Description: Biomicroscopy is analyzed for hema-copolymer and etafilcon A at 1 week. (Scale 0-4, 0=normal, 4=severe).
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
units on a scale
  Conjunctival hyperaemia | 0.96 (0.18) | 0.96 (0.19)
  Limbal hyperameia | 0.86 (0.27) | 0.79 (0.25)
  Corneal vascularisation: number analyzed (Participants) | 29 | 19
  Corneal vascularisation | 0.10 (0.22) | 0.11 (0.26)
  Microcysts | 0.00 (0.00) | 0.00 (0.00)
  Oedema | 0.00 (0.00) | 0.00 (0.00)
  Corenal Staining | 0.26 (0.41) | 0.44 (0.55)
  Conjunctival Staining | 0.37 (0.28) | 0.33 (0.34)
  Papillary Conjunctivitis | 0.87 (0.35) | 0.84 (0.37)

4. Primary Outcome: Lens Surface - Deposition - Hema-copolymer and Etafilcon A
Description: Lens surface of deposition for hema-copolymer and etafilcon A pair of lenses assessed at baseline. (Each pair of lenses worn by the participant was assigned a single grade). Overall score measured by Grade 0-4; 0=absent, clean surface, 4= multiple deposits.
Time Frame: Baseline
Population: All 30 subjects were dispensed lenses, and lens surface of deposition measurements were obtained at baseline.
Measure: Number; unit: participants
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 30 | 30
participants
  Grade 0 | 29 | 30
  Grade 1 | 1 | 0
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

5. Primary Outcome: Lens Surface - Deposition - Hema-copolymer and Etafilcon A
Description: Lens surface of deposition for hema-copolymer and etafilcon A pair of lenses assessed at 1 week. (Each pair of lenses worn by the participant was assigned a single grade). Overall score measured by Grade 0-4; 0=absent, clean surface, 4= multiple deposits.
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Number; unit: participants
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
participants
  Grade 0 | 26 | 14
  Grade 1 | 3 | 6
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

6. Primary Outcome: Lens Surface - Debris - Hema-copolymer and Etafilcon A
Description: Lens surface of debris for hema-copolymer and etafilcon A pair of lenses assessed at baseline. (Each pair of lenses worn by the participant was assigned a single grade). Overall score measured by Grade 0-4; 0=no debris present, 4=debris present more than two thirds of area beneath lens.
Time Frame: Baseline
Population: All 30 subjects were dispensed lenses, and lens surface of debris measurements were obtained at baseline.
Measure: Number; unit: participants
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 30 | 30
participants
  Grade 0 | 28 | 27
  Grade 1 | 1 | 3
  Grade 2 | 1 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

7. Primary Outcome: Lens Surface - Debris - Hema-copolymer and Etafilcon A
Description: Lens surface of debris for hema-copolymer and etafilcon A pair of lenses assessed at 1 week. (Each pair of lenses worn by the participant was assigned a single grade). Overall score measured by Grade 0-4; 0=no debris present, 4=debris present more than two thirds of area beneath lens.
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Number; unit: participants
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
participants
  Grade 0 | 29 | 18
  Grade 1 | 0 | 2
  Grade 2 | 0 | 0
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

8. Primary Outcome: Lens Surface - Wettability - Hema-copolymer and Etafilcon A
Description: Lens surface of wettability for hema-copolymer and etafilcon A pair of lenses assessed at baseline. (Each pair of lenses worn by the participant was assigned a single grade). Overall score measured by Grade 0-4; 0=fully wetting lens surface, 4=presence of one or more non-wetting areas.
Time Frame: Baseline
Population: All 30 subjects were dispensed lenses, and lens surface of wettability measurements were obtained at baseline.
Measure: Number; unit: participants
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 30 | 30
participants
  Grade 0 | 27 | 25
  Grade 1 | 2 | 4
  Grade 2 | 1 | 1
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

9. Primary Outcome: Lens Surface - Wettability - Hema-copolymer and Etafilcon A
Description: Lens surface of wettability for hema-copolymer and etafilcon A pair lenses assessed at 1 week. (Each pair of lenses worn by the participant was assigned a single grade). Overall score measured by Grade 0-4; 0=fully wetting lens surface, 4=presence of one or more non-wetting areas.
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Number; unit: participants
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
participants
  Grade 0 | 19 | 13
  Grade 1 | 6 | 6
  Grade 2 | 4 | 1
  Grade 3 | 0 | 0
  Grade 4 | 0 | 0

10. Primary Outcome: Lens Fit - Horizontal Centration - Hema-copolymer and Etafilcon A
Description: Lens fit of horizontal centration for hema-copolymer and etafilcon A lenses assessed at baseline. Overall score measured by extremely nasal, slightly nasal, optimum, slightly temporal, extremely temporal
Time Frame: Baseline
Population: All 30 subjects were dispensed lenses, and lens fit of horizontal centration measurements were obtained at baseline.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 30 | 30
Number analyzed (Eyes) | 60 | 60
Eyes
  Extremely Nasal | 0 | 0
  Slightly Nasal | 1 | 1
  Optimum | 21 | 19
  Slightly Temporal | 38 | 40
  Extremely Temporal | 0 | 0

11. Primary Outcome: Lens Fit - Horizontal Centration - Hema-copolymer and Etafilcon A
Description: Lens fit of horizontal centration for hema-copolymer and etafilcon A lenses assessed at 1 week. Overall score measured by extremely nasal, slightly nasal, optimum, slightly temporal, extremely temporal
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
Number analyzed (Eyes) | 58 | 40
Eyes
  Extremely Nasal | 0 | 0
  Slightly Nasal | 2 | 0
  Optimum | 11 | 13
  Slightly Temporal | 45 | 27
  Extremely Temporal | 0 | 0

12. Primary Outcome: Lens Fit - Vertical Centration - Hema-copolymer and Etafilcon A
Description: Lens fit of vertical centration for hema-copolymer and etafilcon A lenses assessed at baseline. Overall score measured by extremely inferior, slightly inferior, optimum, slightly superior, extremely superior
Time Frame: Baseline
Population: All 30 subjects were dispensed lenses, and lens fit of vertical centration measurements were obtained at baseline.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 30 | 30
Number analyzed (Eyes) | 60 | 60
Eyes
  Extremely Inferior | 0 | 2
  Slightly Inferior | 22 | 24
  Optimum | 28 | 19
  Slightly Superior | 10 | 15
  Extremely Superior | 0 | 0

13. Primary Outcome: Lens Fit - Vertical Centration - Hema-copolymer and Etafilcon A
Description: Lens fit of vertical centration for hema-copolymer and etafilcon A lenses assessed at 1 week. Overall score measured by extremely inferior, slightly inferior, optimum, slightly superior, extremely superior
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
Number analyzed (Eyes) | 58 | 40
Eyes
  Extremely Inferior | 0 | 0
  Slightly Inferior | 35 | 11
  Optimum | 16 | 17
  Slightly Superior | 7 | 12
  Extremely Superior | 0 | 0

14. Primary Outcome: Lens Fit - Corneal Centration - Hema-copolymer and Etafilcon A
Description: Lens fit of corneal centration for hema-copolymer and etafilcon A lenses assessed at baseline. Overall score measured by extremely inadequate, slightly inadequate, optimum, slightly excessive, extremely excessive
Time Frame: Baseline
Population: All 30 subjects were dispensed lenses, and lens fit of corneal centration measurements were obtained at baseline.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 30 | 30
Number analyzed (Eyes) | 60 | 60
Eyes
  Extremely Inadequate | 0 | 6
  Slightly Inadequate | 1 | 8
  Optimum | 57 | 46
  Slightly Excessive | 2 | 0
  Extremely Excessive | 0 | 0

15. Primary Outcome: Lens Fit - Corneal Centration - Hema-copolymer and Etafilcon A
Description: Lens fit of corneal centration for hema-copolymer and etafilcon A lenses assessed at 1 week. Overall score measured by extremely inadequate, slightly inadequate, optimum, slightly excessive, extremely excessive
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
Number analyzed (Eyes) | 58 | 40
Eyes
  Extremely Inadequate | 0 | 0
  Slightly Inadequate | 3 | 0
  Optimum | 53 | 40
  Slightly Excessive | 2 | 0
  Extremely Excessive | 0 | 0

16. Primary Outcome: Lens Fit - Lens Movement - Hema-copolymer and Etafilcon A
Description: Lens fit of lens movement for hema-copolymer and etafilcon A lenses assessed at baseline. Overall score measured by extremely inadequate, slightly inadequate, optimum, slightly excessive, extremely excessive
Time Frame: Baseline
Population: All 30 subjects were dispensed lenses, and lens movement measurements were obtained at baseline.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 30 | 30
Number analyzed (Eyes) | 60 | 60
Eyes
  Extremely Inadequate | 0 | 0
  Slightly Inadequate | 7 | 0
  Optimum | 41 | 35
  Slightly Excessive | 12 | 16
  Extremely Excessive | 0 | 9

17. Primary Outcome: Lens Fit - Lens Movement - Hema-copolymer and Etafilcon A
Description: Lens fit of lens movement for hema-copolymer and etafilcon A lenses assessed at 1 week. Overall score measured by extremely inadequate, slightly inadequate, optimum, slightly excessive, extremely excessive
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
Number analyzed (Eyes) | 58 | 40
Eyes
  Extremely Inadequate | 0 | 0
  Slightly Inadequate | 5 | 2
  Optimum | 33 | 28
  Slightly Excessive | 20 | 8
  Extremely Excessive | 0 | 2

18. Primary Outcome: Comfort Preference (Subjective Assessment) - Hema-copolymer and Etafilcon A
Description: Subjective Assessment of comfort preference for hema-copolymer and etafilcon A assessed at baseline. Scale 0-100, 0=causes pain, 100= excellent.
Time Frame: Baseline
Population: 7 subjects discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 24
units on a scale | 82.2 (13.6) | 84.5 (15.3)

19. Primary Outcome: Comfort Preference (Subjective Assessment) - Hema-copolymer and Etafilcon A
Description: Subjective Assessment of comfort preference after insertion and before removal for hema-copolymer and etafilcon A lenses is assessed at 1 week. Scale 0-100, 0=causes pain, 100= excellent.
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
units on a scale
  Comfort after insertion | 80.8 (17.0) | 76.0 (16.1)
  Comfort before removal | 69.1 (19.2) | 66.6 (19.5)
  Overall comfort | 75.8 (16.5) | 69.5 (20.8)

20. Primary Outcome: Vision Preference (Subjective Assessment) - Hema-copolymer and Etafilcon A
Description: Subjective Assessment of vision preference for hema-copolymer and etafilcon A lenses assessed at baseline. Scale 0-100, 0=unacceptable, 100= excellent.
Time Frame: Baseline
Population: 8 subjects discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 23
units on a scale | 87.6 (11.5) | 84.4 (12.3)

21. Primary Outcome: Vision Preference (Subjective Assessment) - Hema-copolymer and Etafilcon A
Description: Subjective Assessment of vision preference for hema-copolymer and etafilcon A lenses assessed at 1 week. Scale 0-100, 0=unacceptable, 100= excellent.
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
units on a scale
  Distance vision | 85.6 (11.3) | 71.6 (22.7)
  Vision at night | 83.3 (14.0) | 65.0 (21.3)
  Variable vision | 83.1 (17.4) | 67.4 (22.7)

22. Primary Outcome: Peripheral Blur (Subjective Assessment) - Hema-copolymer and Etafilcon A
Description: Subjective Assessment of peripheral blur is assessed at baseline. Scale 0-100, 0=unacceptable, 100= excellent.
Time Frame: Baseline
Population: 8 subjects discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 23
units on a scale | 85.1 (14.7) | 87.6 (14.9)

23. Primary Outcome: Peripheral Blur (Subjective Assessment) - Hema-copolymer and Etafilcon A
Description: Subjective Assessment of peripheral blur assessed at 1 week. Scale 0-100, 0=unacceptable, 100= excellent.
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
units on a scale | 80.2 (16.4) | 76.4 (17.3)

24. Primary Outcome: Ocular Redness (Subjective Assessment) - Hema-copolymer and Etafilcon A
Description: Subjective Assessment of ocular redness for hema-copolymer and etafilcon A lenses lenses assessed at 1 week. Scale 0-100, 0=extremely poor, 100= excellent.
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
units on a scale | 87.2 (15.7) | 89.0 (9.0)

25. Primary Outcome: Handling (Subjective Assessment) - Hema-copolymer and Etafilcon A
Description: Subjective Assessment of handling (ease of insertion and ease of removal) for hema-copolymer and etafilcon A lenses assessed at 1 week. Scale 0-100, 0=unmanageable, 100= excellent.
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
units on a scale
  Ease of insertion | 92.0 (10.3) | 77.5 (18.2)
  Ease of removal | 95.2 (8.1) | 90.5 (18.3)

26. Primary Outcome: Attractiveness (Subjective Assessment) - Hema-copolymer and Etafilcon A
Description: Subjective Assessment of attractiveness for hema-copolymer and etafilcon A lenses assessed at baseline. Scale 0-100, 0=extremely poor, 100= excellent.
Time Frame: Baseline
Population: 8 subjects discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 23
units on a scale | 66.9 (16.5) | 67.4 (16.7)

27. Primary Outcome: Attractiveness (Subjective Assessment) - Hema-copolymer and Etafilcon A
Description: Subjective Assessment of attractiveness for hema-copolymer and etafilcon A lenses assessed at 1 week. Scale 0-100, 0=extremely poor, 100= excellent.
Time Frame: 1 week
Population: 11 subjects discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 20
units on a scale | 66.7 (20.0) | 68.0 (20.2)

28. Primary Outcome: Overall Impression (Subjective Assessment) - Hema-copolymer and Etafilcon A
Description: Subjective assessment of the overall impression for hema-copolymer and etafilcon A lenses assessed at baseline. Scale 0-100, 0=extremely poor, 100= excellent.
Time Frame: Baseline
Population: 8 subjects discontinued the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 29 | 23
units on a scale | 81.3 (14.6) | 78.9 (14.5)

29. Primary Outcome: Overall Impression (Subjective Assessment) - Hema-copolymer and Etafilcon A
Description: Subjective assessment of the overall impression for hema-copolymer and etafilcon A lenses assessed at 1 week. Scale 0-100, 0=extremely poor, 100= excellent.
Time Frame: 1 week
Population: 11 subjects discontinued the study. Missing data of 1 subject for hema-copolymer group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Number analyzed (Participants) | 28 | 20
units on a scale | 75.0 (15.2) | 63.9 (21.5)

ADVERSE EVENTS:
Arm/Group | Hema-copolymer Lens | Etafilcon A Lens
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 1/19 | 0/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hema-copolymer Lens (N=19) | Etafilcon A Lens (N=19)
Unilateral red eye (Eye disorders) | 1 (1) | 0 (0) — Unilateral red eye on removal of the hema-copolymer lens. Symptoms resolved overnight and normal wear was resumed the next day.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor that restricts the PI's right to discuss or publish trial results after the trial is completed without prior approval of Sponsor.

The investigator will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.